CLINICAL TRIAL: NCT03247049
Title: Predicting Long Term Survival in Patients With Primary Intracerebral Hemorrhage. Development and Validation of the ICHCat in Primary Care.
Brief Title: Prognosis in Intracerebral Hemorrhage. The ICHCat Score in Primary Care.
Acronym: ICHCat
Status: Completed | Type: Observational
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Josep Lluís Clua Espuny, PhD, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Other Study IDs: IDIAP Jordi Gol code P16/087
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Intracerebral Hemorrhage; Outcome; Survival; Primary Care; Hazard Risk
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The clinical evidence shows that patients with a first episode of intracerebral hemorrhage (ICH) are increasingly old and with greater comorbidity with a recognized impact over mortality. The prediction of the outcome of ICH is not only crucial in the emergin attention to identify those patients with favorable criteria that can benefit from possible treatments; but also after hospital discharge, in primary care where the prediction should facilitate the organization and management of a wide variety of resources: familiar, health and social welfare. Even though there are different scales that predict mortality, these are not sufficiently useful in choosing a treatment or do not provide sufficient data to the family to decide.

Due to the characteristics of the population with ICH described in these works, it seems useful to propose a prognostic index (ICHCat) to identify the variables associated to its incidence and mortality and that, in addition, to make adjustments in the comparisons of the survival between different series of patients or different treatment modalities in primary care.

DETAILED DESCRIPTION:
The authors carried out a multicentric and retrospective study of a cohort with an episode of ICH in the period between 2006-2016. The objective of this phase is to design a predictive index (ICHCat) of mortality in patients with an episode of ICH. Patient outcome was followed until death all causes or study end (30.09.2016) since date of ICH in the electronic health record. All people included were managed by the Public Health System in Catalonia. Registry information was collected from the government-run healthcare provider responsible for all inpatient care in the county.

Predictor Variables

Predictor variables were considered if they were viewed as commonly measured and available in primary care and with potential evidence of an association with ICH risk. Candidate variables included:

Sex: woman (0) man (1) Age: <80 year-old (1), ≥80 year-old (2). Number CCP criteria: <4 (0) ≥4 (1). Charlson comorbidity index. Short version. Current medications were asked about during the home visit and confirmed in medical records. Polypharmacy (defined as five or more daily medications): <5 (0), between 5-9 (1), and ≥10 (2). Oral anticoagulants (acenocumarol or warfarin) with TTR ≥60% (1), if TRT <60% (2) or New Oral Anticoagulants NOACs (0). Antidepressants and/or, sedating or other drugs affecting the neurologic system: man (1), woman (2). If there was a diagnostic of "atrial fibrillation", CHA2DS2VASC and HAS-BLED scores were included.

Recurrent falls or fall risk: no (0), yes (1). Hypertension not controlled by therapy (≥ 160/90 mmHg): no (0), yes (1). BP was measured as an average of separated follow-up measurements last six months.

Alcoholism abuse vs dependence: no (0), yes (1) Presence de cognitive impairment: a disease-specific diagnosis of cognitive impairment and/or prescription of specific treatment, without specification of sub-type or severity, was used and mesured by Pfeiffer test [2]: [0-2 errors] = Intact Intellectual Functioning (1); [≥3 errors] = Mild to severe Intellectual Impairment (2)].

Presence de disability: score in [Barthel ≥60 (1) <60 (2)] or in [Rankin <4 (1) 5(2)] were used to assess dependence in ADL Functional status: (0) Autonomus (1) Residual with caretaker (2) Dependence with caretaker (3) Long stay

Socio familiar risk: score in Gijon[18] scale 10-14 (1) ≥15 (2)]

Primary Outcome Given the limited survival, the primary outcome was death all causes occurring within the 5-year follow-up after the ICH episode.

Predictions of ICH mortality risk were based on Cox proportional-hazards regression models. All potential predictors were considered in a multivariate logistic regression, and a backward step selection procedure was carried out to pick the variables that composed the best model. Subsequently design a predictive model of multivariate Cox regression analysis to define the weight of each of the pathologies in the mortality. To assign the weight according to the value HR took into account only those with a HR ≥1.2 in the multivariate model approximating the value of HR to the nearest whole number:

* HR between 1.20 and 1.49 scored with 1.
* HR between 1.50 and 2.49 with 2.
* HR between 2.50 and 3.49 received 3, and so on.

The final score for each patient (ICH) was made up of the sum of their scores by age and comorbidity. To check the validity of the index we define the following levels of mortality risk:

* Low risk: 0-1 points.
* Medium Risk: from 2 to 5 points.
* High Risk: of 6 or more points.

The authors estimate the survival probability of each risk group according to the Kaplan-Meier method and compared these curves using the Log-Rank test. It will be used ROC curves i the AUC to assess the ability of the index ICH to perform properly the assignment of patients to different risk groups. The hazard ratio according to the proportional hazards model categorized in their levels of risk, in order to observe the increase in the risk of death that occurs from a risk group to the next. The statistical analysis consisted of a multivariate logistic regression model. The model selection has been caried out with an AIC-led forward step selection method. To ensure internal validity, 20% of data has been discarded in the phase of constructing the model and only used to assess model performance using ROC curves and the AUC.

In a second phase, there will be a retrospective study of validation in the cohort of patients PCC of the territory with an episode of ICH.

ELIGIBILITY:
Inclusion Criteria:

* Have been suffered a Intracranial Hemorrhage

Exclusion Criteria:

* <15 and >90 year-old

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort with an episode of ICH in the period April 1, 2006 to Setember 30, 2016.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Death all causes | Within 5 years follow-up after episode ICH
  Death all causes

CONTACTS AND LOCATIONS:
Overall Officials: V Francisco Gil-Guillen, PhD, Study Chair — Universidad Miguel Hernandez

IPD SHARING:
Plan to Share IPD: Undecided
All IPD will be shared after definitive validation

REFERENCES:
- [Result] Gonzalez-Henares A, Clua-Espuny JL, Gil-Guillen VF, Panisello-Tafalla A, Queralt-Tomas ML, Ripolles-Vicente R, Lopez-Pablo C, Lucas-Noll J, Equipo de Investigacion Ebrictus Ede I. [Incidence and preventability of haemorrhagic strokes. Results of the Ebrictus register]. Rev Neurol. 2016 May 1;62(9):385-95. Spanish. PMID 27113062
- [Derived] Lorman-Carbo B, Clua-Espuny JL, Muria-Subirats E, Ballesta-Ors J, Gonzalez-Henares MA, Fernandez-Saez J, Martin-Lujan FM; on behalf Ebrictus Research Group. Complex chronic patients as an emergent group with high risk of intracerebral haemorrhage: an observational cohort study. BMC Geriatr. 2021 Feb 5;21(1):106. doi: 10.1186/s12877-021-02004-4. PMID 33546615
- [Derived] Gonzalez-Henares MA, Clua-Espuny JL, Lorman-Carbo B, Fernandez-Saez J, Queralt-Tomas L, Muria-Subirats E, Ballesta-Ors J, Gil-Guillen JV. Risk of Long-Term Mortality for Complex Chronic Patients with Intracerebral Hemorrhage: A Population-Based e-Cohort Observational Study. Adv Ther. 2020 Feb;37(2):833-846. doi: 10.1007/s12325-019-01206-y. Epub 2019 Dec 26. PMID 31879838